CLINICAL TRIAL: NCT04849689
Title: Whole-Food, Plant-Based Lifestyle Program Preserves Muscle Mass During Body Mass/Fat Mass Loss
Brief Title: WFPB Lifestyle and Muscle Mass Preservation
Acronym: WFPBmuscle
Status: Completed | Type: Observational
Sponsor: Barbara Jakše s.p. (Other)
Responsible Party: Principal Investigator, Boštjan Jakše, Principal Investigator, Barbara Jakše s.p.
Other Study IDs: KR5
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Body Weight; Body Image; Body Weight Changes; Muscle Loss
Keywords: Body composition; Plant-based diet; Lifestyle; Physical activity; Support system; Muscle mass preservation; Fat loss
MeSH Terms: conditions — Body Weight; Body Weight Changes; Muscular Atrophy; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

INTERVENTIONS:
Behavioral: Whole-food, plant-based lifestyle — The WFPB lifestyle program included:
  1. Nutrition/plant-based food (energy intake: at least 90% of whole-food, plant-based diet and ≤ 10% of energy intake from plant-based meal replacements (PBMR) and dietary supplements (e.g., vitamin B12, D, and EPA and DHA omega-3 fatty acids).
  2. Physical activity (habitual; organized and other).
  3. Support system (lectures, workshops and individual nutrition counselling, grocery shopping assistance, cooking classes, regular measurements body composition, food logging, regular medical monitoring).

SUMMARY:
Body fat (BF) and muscle mass showed opposing association with mortality. Whole-food, plant-based (WFPB) lifestyle programs has been on the rise lately especially due to impressive health benefits.

The results of research on the effectiveness of popular weight loss diets in obese subjects showed 20 to 30% loss of lean muscle mass within to the total body weight loss, whereas in the whole-food, plant-based (vegan) diet the loss was up to 42%.

Therefore, an open research problem is to find a way how to improve body composition in an effective and healthy way (i.e., losing of excess BF while maintaining muscle mass as much as possible) but still using stric plant-based (vegan) diet.

Investigators will perform retrospective analysis of measurements of body composition and phase angle values of aprox. 200 participants who were on a WFPB lifestyle program from 2016 to 2021 and performed two successive measurements (initial and follow up (FU)), without body mass index (BMI) limitation on same medically approved and calibrated bioelectrical impedance (Tanita 780 S MA, Tokyo, Japan) and were not yet included in our previous studies. A WFPB lifestyle program were consisted of nutrition (i), (ii) physical activity and (iii) support system.

Primary outcome include the following measures: BF % and FFM and to examine the change from initial values to FU values (by gender), according BMI classification (e.g,, normal, pre-obese and obese) with subanalysis for those participants who lost up to 5 kg/more and those who lost 5 kg or more of body weight.

DETAILED DESCRIPTION:
Many people are increasingly using a variety of dietary practices to manage overweight and obesity. Many people are increasingly using a variety of dietary practices to manage overweight and obesity.

Investigators will investigate the muscle mass preservation of participants on our 12-year lasting ongoing, community-based (free-living), WFPB lifestyle program during the weight/fat loss of participants.

The primary outcome is the BF %, and FFM change from initial values to FU values (for whole sample and by gender).

Secondary outcome include correlation between BMI, BF % and FFM, and PhA. Based on our experiences we believe that some participants that follow our WFPB lifestyle program may initially "afraid" to eat, according to the instructions, each meal to satiety (ad libitum). The reason lies in the typical weight loss recommendation in Western-type lifestyle that advise "eating less".

The body composition measures will include body height (BH; measured via standardized medical approved professional personal floor scale with stand (Kern, MPE 250K100HM, Kern & Sohn, Balingen, Germany), body mass (BM), BF mass and BF %, FFM, bone mineral mass (BMM), visceral fat (VF), total body water (TBW), extracellular water (ECW), intracellular water (ICW), the ratio, whole body phase angle (PhA), all via medically approved and calibrated bioelectrical impedance Tanita 780 S MA (Tanita Corporation, Tokyo, Japan) and the use of corresponding protocols (e.g., for BMI).

ELIGIBILITY:
Inclusion Criteria:

* Using WFPB lifestyle program.
* Were measured on a body composition analyzer at least two successive times on the same body composition montor Tanita 780 S MA, Tokyo, Japan (at baseline, follow up) in a row at different intervals (i.e., before the start of the program and as part of follow up).
* Follow up up to 6 months
* Baseline BMI status was not an exclusion criteria.
* Data of participants that did not participate yet in our previous research.
* No medication use

If the individual performed more than two consecutive measurements, only the first two were included in the analysis.

Exclusion Criteria:

* Being on vegan diet before joined in our program.
* Being adult (e.g., older than 18-years) before the start of the program.
* Participating in our preivous research using WFPB lifestyle program.
* Without severe chronic diseases or physical limitations (described bellow).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will examine the body composition data of healthy adults from Slovenia (European Union) that were without preference toward plant-based diet before entering to the program. As healthy adults we mean that used data were from participants without serious comorbidities (i.e., having autoimmune or neurodegenerative disorders), physical limitations or taking medicine (for blood pressure, blood sugar or cholesterol).
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Fat- free mass (FFM) change | Baseline, up to 6 months
  Muscle mass measured with bioimpedance analysis
Body fat mass percentage (BF %) change | Baseline, up to 6 months
  Fat mass measured with bioimpedance analysis
Body mass index (BMI) change | Baseline, up to 6 months
  Body mass index measured with bioimpedance analysis

SECONDARY OUTCOMES:
Correlation between BMI, BF % and FFM and phase angle | Baseline, up to 6 months
  Correlation status of variables

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Pinter, PhD, Study Chair — University of Ljubljana; Bostjan Jakse, PhD student, Principal Investigator — University of Ljubljana
Locations (1):
- PDP Spodnje Črnuče, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finucane MM, Stevens GA, Cowan MJ, Danaei G, Lin JK, Paciorek CJ, Singh GM, Gutierrez HR, Lu Y, Bahalim AN, Farzadfar F, Riley LM, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Body Mass Index). National, regional, and global trends in body-mass index since 1980: systematic analysis of health examination surveys and epidemiological studies with 960 country-years and 9.1 million participants. Lancet. 2011 Feb 12;377(9765):557-67. doi: 10.1016/S0140-6736(10)62037-5. Epub 2011 Feb 3. PMID 21295846
- [Background] Turner-McGrievy GM, Barnard ND, Cohen J, Jenkins DJ, Gloede L, Green AA. Changes in nutrient intake and dietary quality among participants with type 2 diabetes following a low-fat vegan diet or a conventional diabetes diet for 22 weeks. J Am Diet Assoc. 2008 Oct;108(10):1636-45. doi: 10.1016/j.jada.2008.07.015. PMID 18926128
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Kent L, Morton D, Hurlow T, Rankin P, Hanna A, Diehl H. Long-term effectiveness of the community-based Complete Health Improvement Program (CHIP) lifestyle intervention: a cohort study. BMJ Open. 2013 Nov 20;3(11):e003751. doi: 10.1136/bmjopen-2013-003751. PMID 24259389
- [Background] Johns DJ, Hartmann-Boyce J, Jebb SA, Aveyard P; Behavioural Weight Management Review Group. Diet or exercise interventions vs combined behavioral weight management programs: a systematic review and meta-analysis of direct comparisons. J Acad Nutr Diet. 2014 Oct;114(10):1557-68. doi: 10.1016/j.jand.2014.07.005. PMID 25257365
- [Background] Cava E, Yeat NC, Mittendorfer B. Preserving Healthy Muscle during Weight Loss. Adv Nutr. 2017 May 15;8(3):511-519. doi: 10.3945/an.116.014506. Print 2017 May. PMID 28507015